CLINICAL TRIAL: NCT01349972
Title: Randomized Phase II Trial of Timed Sequential Therapy (TST) With Alvocidib (Flavopiridol), Ara-C and Mitoxantrone (FLAM) vs. "7+3" for Adults Age 70 and Under With Newly Diagnosed Acute Myelogenous Leukemia (AML)
Brief Title: Alvocidib, Cytarabine, and Mitoxantrone Hydrochloride or Cytarabine and Daunorubicin Hydrochloride in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02587; NCI-2011-02587 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JHOC-J1101; CDR0000699421; J1101 (Other: Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center); 8972 (Other: CTEP); U01CA070095 (NIH); N01CM00100 (NIH); P30CA006973 (NIH); NCT01413880 (obsolete NCT alias)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — alvocidib; Daunorubicin; Mitoxantrone; Cytarabine

ARMS (2):
- Arm I (alvocidib, cytarabine, mitoxantrone hydrochloride) (Experimental): Patients receive alvocidib IV over 1 hour on days 1-3, cytarabine IV over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9. Patients who achieve complete or partial response to the first course (completion of all doses) may receive a second course of treatment or high-dose cytarabine after 21-63 days following blood count recovery, and/or undergo allogeneic bone marrow transplant.
  Interventions: Drug: alvocidib; Drug: mitoxantrone hydrochloride; Drug: cytarabine
- Arm II (cytarabine, daunorubicin hydrochloride) (Active Comparator): Patients receive cytarabine IV continuously on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients who have residual disease on day 14 may receive additional cytarabine for 5 days and daunorubicin hydrochloride for 2 days.
  Interventions: Drug: daunorubicin hydrochloride; Drug: cytarabine

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
  Arms: Arm I (alvocidib, cytarabine, mitoxantrone hydrochloride)
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
  Arms: Arm II (cytarabine, daunorubicin hydrochloride)
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ
  Arms: Arm I (alvocidib, cytarabine, mitoxantrone hydrochloride)
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This randomized phase II trial is studying how alvocidib, cytarabine, and mitoxantrone hydrochloride work compared to cytarabine and daunorubicin hydrochloride in treating patients with newly diagnosed acute myeloid leukemia. Alvocidib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine, mitoxantrone hydrochloride, and daunorubicin hydrochloride work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving alvocidib, cytarabine, and mitoxantrone hydrochloride is more effective than giving cytarabine and daunorubicin hydrochloride in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rate of complete remission (CR) after 1 course of induction therapy with the timed-sequential combination of alvocidib (flavopiridol), cytarabine (cytosine arabinoside [ara-C]), and mitoxantrone hydrochloride (FLAM) vs traditional "7+3" cytarabine and daunorubicin hydrochloride (ara-C + Daunorubicin) for adults (age 18 to 70) with newly diagnosed, previously untreated, intermediate-risk or poor-risk acute myelogenous leukemia (AML).

SECONDARY OBJECTIVES:

I. To evaluate and compare the toxicities of FLAM vs 7+3. II. To compare the 2-year disease-free survival (DFS) and overall survival (OS) in response to FLAM vs 7+3.

III. To detect and compare the presence of minimal-residual disease (MRD) remaining after FLAM vs 7+3.

IV. To determine the expression of ABC transport proteins multidrug resistance 1 (MDR1, ABCB1) and breast cancer resistance protein (BCRP, ABCG2) on AML blasts pretreatment and correlate the expressions of one or both proteins with CR and DFS in response to FLAM vs 7+3.

OUTLINE: This is a multicenter study. Patients are stratified according to risk features: age (< 50 vs >= 50), secondary AML (pre-existing myelodysplatic syndrome [MDS], myeloproliferative diseases [MPD], treatment-related [t]-AML, or severe multi-lineage dysplasia) and/or known adverse cytogenetics, and hyperleukocytosis (white blood cells [WBC] >= 50,000/mm^3). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive alvocidib intravenously (IV) over 1 hour on days 1-3, cytarabine IV over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9. Patients who achieve complete or partial response to the first course (completion of all doses) may receive a second course of treatment or high-dose cytarabine after 21-63 days following blood count recovery, and/or undergo allogeneic bone marrow transplant.

ARM II: Patients receive cytarabine IV continuously on days 1-7 and daunorubicin hydrochloride IV on days 1-3. Patients who have residual disease on day 14 may receive additional cytarabine for 5 days and daunorubicin hydrochloride for 2 days. Patients may undergo blood and bone marrow collection for correlative studies.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All adults with established, pathologically confirmed diagnoses of newly diagnosed AML and adults with newly diagnosed AML, excluding newly diagnosed core-binding factor (CBF) AMLs and acute progranulocytic leukemia (APL, M3), will be considered eligible for study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3

  * Patients >= 65 years of age must have ECOG PS =< 2 prior to developing leukemic symptoms
* Serum creatinine ≤ 2.0 mg/dL
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 5 times upper limit of normal (ULN) (unless leukemic infiltration)
* Total bilirubin =< 2.0 mg/dL (unless Gilbert disease, hemolysis, or leukemia)
* Left ventricular ejection fraction ≥ 45%
* Newly diagnosed AML, subtypes M0, 1, 2, 4-7 but excluding M3 (APL), including those with the following poor risk features:

  * Antecedent hematologic disorder including myelodysplasia (MDS)-related AML (MDS/AML) and prior myeloproliferative disorder (MPD)
  * Treatment-related myeloid neoplasms (t-AML/t-MDS)
  * Myeloid sarcoma, myeloid proliferations related to Down Syndrome, and blastic plasmacytoid dendritic cell neoplasm
  * AML with multilineage dysplasia (AML-MLD)
  * Adverse cytogenetics (defined as -5/-5q; -7/-7q; abnormal 3q, 9q, 11q, 20q, 21q, or 17p; t(6;9); t(9;22); trisomy 8; trisomy 13; trisomy 21; and complex karyotypes (≥ 3 unrelated abnormalities)
* Patients who have received hydroxyurea alone or have received non-cytotoxic therapies previously for myelodysplasia (MDS) or myeloproliferative disorder (MPD) (e.g., thalidomide or lenalidomide, interferon, cytokines, 5-azacytidine or decitabine, histone deacetylase inhibitors, low-dose cyclophosphamide [cytoxan], tyrosine kinase [TK] or dual TK/src inhibitors) will be eligible for this trial

  * At least 24 hours since prior leukopheresis or hydroxyurea for cytoreduction

Exclusion Criteria:

* Any previous treatment with flavopiridol
* Concomitant chemotherapy, radiation therapy, or immunotherapy
* Hyperleukocytosis with >= 50,000 blasts/uL; leukopheresis or hydroxyurea may be used immediately prior to study drug administration for cytoreduction; must be stopped 24 hours before first dose of study chemotherapy
* CBF AMLs associated with t(8;21) or M4eo subtype (inv[16] or t[16;16]), as diagnosed by morphologic criteria, flow cytometric characteristics, and rapid cytogenetics or FISH or molecular testing
* Acute Progranulocytic Leukemia (APL, M3)
* Active central nervous system (CNS) leukemia
* Active, uncontrolled infection; patients with infection under active treatment and controlled with antibiotics are eligible
* Active, uncontrolled graft vs. host disease (GVHD) following allogeneic transplant for non-AML condition (e.g. MDS, lymphoid malignancy, aplastic anemia); patients with GVHD controlled on stable doses of immunosuppressants are eligible
* Presence of other life-threatening illness
* Patients with mental deficits and/or psychiatric history that preclude them form giving informed consent or from following protocol
* Pregnant and nursing patients are excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Smith, Principal Investigator — Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center
Locations (11):
- United States (11):
  - Mayo Clinic Scottsdale-Phoenix, Scottsdale, Arizona
  - Moffitt Cancer Center, Tampa, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Zeidner JF, Foster MC, Blackford AL, Litzow MR, Morris LE, Strickland SA, Lancet JE, Bose P, Levy MY, Tibes R, Gojo I, Gocke CD, Rosner GL, Little RF, Wright JJ, Doyle LA, Smith BD, Karp JE. Randomized multicenter phase II study of flavopiridol (alvocidib), cytarabine, and mitoxantrone (FLAM) versus cytarabine/daunorubicin (7+3) in newly diagnosed acute myeloid leukemia. Haematologica. 2015 Sep;100(9):1172-9. doi: 10.3324/haematol.2015.125849. Epub 2015 May 28. PMID 26022709
- [Derived] Gerber JM, Zeidner JF, Morse S, Blackford AL, Perkins B, Yanagisawa B, Zhang H, Morsberger L, Karp J, Ning Y, Gocke CD, Rosner GL, Smith BD, Jones RJ. Association of acute myeloid leukemia's most immature phenotype with risk groups and outcomes. Haematologica. 2016 May;101(5):607-16. doi: 10.3324/haematol.2015.135194. Epub 2016 Jan 27. PMID 26819054
- See also: Pubmed — http://www.ncbi.nlm.nih.gov/m/pubmed/26022709/?i=1&from=zeidner%20jf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Started | 114 | 58
Completed | 109 | 56
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride) | Total
Number analyzed (Participants) | 114 | 58 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 43 | 122
  >=65 years | 35 | 15 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 27 | 80
  Male | 61 | 31 | 92

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an ANC of at least 1000/cu mm and a platelet count of 100,000/cu mm, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, clearance of disease-associated cytogenetic abnormalities, and clearance of any previously existing extramedullary disease. These criteria are taken from Dohner H, Estey EH, Amadori S, et al. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood 2010;115:453-474
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Number analyzed (Participants) | 109 | 56
participants | 76 | 24

2. Secondary Outcome: Incidence of Toxicities, Characterized by Number of Events by Treatment and Grade
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Time Frame: Up to 14 days after completion of study treatment
Population: Number of evaluable subjects
Measure: Number; unit: Number of events
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Number analyzed (Participants) | 109 | 56
Number of events | 156 | 77

3. Secondary Outcome: Disease-free Survival
Description: Probabilities will be estimated with the Kaplan-Meier estimate. Survival estimates at two years will be estimated. Disease-free survival Overall survival was defined from date of randomization to death or last known follow-up. Event free survival was defined as date of randomization to the first occurrence of persistent AML after 1 cycle of induction, relapse or death. Patients were censored for event free survival if they had received non-protocol therapy or a stem cell transplant.
Time Frame: Time from randomization until death from any cause or relapse or recurrence, assessed up to 2 years
Measure: Median (Full Range); unit: years
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Number analyzed (Participants) | 114 | 58
years | 1.46 [1.06 to 2.11] | 1.85 [1.35 to 3.33]

4. Secondary Outcome: Overall Survival
Description: Probabilities will be estimated with the Kaplan-Meier estimate. Survival estimates at two years will be estimated.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Number analyzed (Participants) | 109 | 56
years | 1.46 [0.09 to 2.12] | 1.850 [1.35 to 3.33]

5. Secondary Outcome: Number of Patients With Minimal Residual Disease
Description: Comparisons of the treatments with respect to MRD will be based on the number of patients with MRD at day 14 after the start of treatment.
Time Frame: From study start to 14 days after the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Number analyzed (Participants) | 102 | 55
Participants | 26 | 24

6. Secondary Outcome: Progression-free Survival
Description: Probabilities will be estimated with the Kaplan-Meier estimate. Survival estimates at two years will be estimated.
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Number analyzed (Participants) | 76 | 26
years | 0.81 [0.42 to 0.98] | 0.28 [0.11 to 1.11]

ADVERSE EVENTS:
Arm/Group | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) | Arm II (Cytarabine, Daunorubicin Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 53/114 | 21/58
Other Adverse Events (participants affected / at risk) | 32/114 | 21/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) (N=114) | Arm II (Cytarabine, Daunorubicin Hydrochloride) (N=58)
bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
cardiac chest pain (Cardiac disorders) | 1 (1) | 0 (0)
heart failure (Cardiac disorders) | 2 (2) | 0 (0)
left ventricular systolic dysfunction (Cardiac disorders) | 5 (5) | 0 (0)
myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
thyrotoxicosis (Endocrine disorders) | 1 (1) | 0 (0)
ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
peritoneal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal hemmorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
death (General disorders) | 1 (1) | 0 (0)
fever (General disorders) | 2 (2) | 0 (0)
cytokine release syndrome (Immune system disorders) | 3 (3) | 2 (2)
appendicitis (Infections and infestations) | 1 (1) | 0 (0)
lung infection (Infections and infestations) | 2 (2) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
sogt tissue infection (Immune system disorders) | 1 (1) | 0 (0)
blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
creatinine increased (Investigations) | 1 (1) | 0 (0)
QTc prolonged (Investigations) | 1 (1) | 0 (0)
alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
tumor lysis syndrome (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
necrotic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
thrombotic event (Vascular disorders) | 1 (1) | 0 (0)
adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Alvocidib, Cytarabine, Mitoxantrone Hydrochloride) (N=114) | Arm II (Cytarabine, Daunorubicin Hydrochloride) (N=58)
Febril eNeutropenia (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Catheter Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Infectious Enterocolitis (Infections and infestations) | 2 (2) | 0 (0)
mucositis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalemia (Investigations) | 1 (1) | 0 (0)
Mypocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Investigations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypocalcemia (Investigations) | 1 (1) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Edema (General disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less